CLINICAL TRIAL: NCT05710887
Title: Inhaled Nitrous Oxide for Acute Suicidality and Depression in the Emergency Department
Brief Title: N2O for Acute Suicidality and Depression in the ED
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB18-1083
Record Dates: First submitted 2023-01-11; First posted 2023-02-02 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Suicidal Ideation; Major Depressive Disorder; Treatment Resistant Depression
Keywords: Suicidal; Depression; Nitrous; Antidepressant; MDD; TRD
MeSH Terms: conditions — Suicidal Ideation; Depressive Disorder, Major; Depressive Disorder, Treatment-Resistant; Depression | interventions — Endothelium-Dependent Relaxing Factors; Inhalation; Nitrous Oxide; salicylhydroxamic acid

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to one of two treatment arms (nitrous vs placebo). Dosing includes a single inhalation session of either 50% Nitrous oxide in oxygen mixture (FiO2 0.5) vs placebo (oxygen-air mixture FiO2 ≈0.3).
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Treatment; Nitrous Oxide 50% (Active Comparator): A single 45-minute session of inhaled 50% nitrous oxide.
  Interventions: Drug: Nitrous oxide gas for inhalation
- Control; Oxygen-air mixture (Placebo Comparator): A single 45-minute session of inhaled Oxygen-air mixture
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nitrous oxide gas for inhalation — Administration of inhaled 50% nitrous oxide in oxygen (FiO2 0.5) will be under the direct supervision of a licensed practitioner who is experienced in the use and administration of the study drug, and is familiar with the indications, effects, dosages, methods, and frequency and duration of administration, and with the hazards, contraindications, and side effects and the precautions to be taken (MD, or CRNA); with study patient monitoring of pulse oximetry, heart rate, respiratory, non-invasive blood pressure, and end-tidal carbon dioxide.
  Other Names: Nitrous Oxide; Nitrous; N2O; Laughing Gas
  Arms: Treatment; Nitrous Oxide 50%
Drug: Placebo — Administration of the placebo (oxygen-air mixture [FiO2 ≈0.3]), will be under the direct supervision of a licensed practitioner who is experienced in the use and administration of the study drug, and is familiar with the indications, effects, dosages, methods, and frequency and duration of administration, and with the hazards, contraindications, and side effects and the precautions to be taken (MD, or CRNA); with study patient monitoring of pulse oximetry, heart rate, respiratory, non-invasive blood pressure, and end-tidal carbon dioxide.
  Other Names: Sham
  Arms: Control; Oxygen-air mixture

SUMMARY:
Investigators are conducting this double-blind, randomized control trial (RCT), to compare inhaled N2O+ treatment as usual (TAU) versus inhaled placebo+TAU; demonstrating the feasibility and tolerability of the intervention in an emergency department (ED) setting on an acutely suicidal population.

DETAILED DESCRIPTION:
Past studies have shown that a single dose of ketamine, an NMDA- receptor antagonist has fast and long lasting anti-depressant effect. Although a promising antidepressant and potential anti-suicidal agent, ketamine has very significant side effects including: dissociation, hallucinations, delusional thinking, cognitive impairment, and significant sympathetic nervous system activation.

Nitrous Oxide (N2O) is an NMDA-receptor antagonist with a well-known safety profile used as an analgesic. In a proof-of-concept pilot study, this study's investigator recently demonstrated that N2O also has rapid and marked antidepressant effects in patients with severe treatment-resistant depression (TRD); further sub-analyses showed N2O significantly reduced suicidal ideation (SI). While N2O administration may lead to a reduction in SI, it remains unknown whether severely suicidal patients requiring hospitalization on inpatient psychiatric units would benefit. Investigators hypothesize that N2O will rapidly and safely dampen suicidal thinking with minimal side effects in this population.

Participants will be randomized to receive either N2O or placebo. The study intervention is in tandem with prescribed treatment-as-usual (TAU) by emergency department physicians relating to diagnosis (depression, anxiety, suicidal ideation); which typically involves anxiolytic medications and/or brief psychotherapy administered by care team psychiatry providers.

Study intervention response will be assessed using a self-administered psychiatric diagnostic tool (Computerized Adaptive Testing Mental Health [CAT-MH] scores relating to suicide, depression, and anxiety; to determine whether a single 45-minute inhalation of nitrous oxide vs placebo reduces symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18-65 years of age, acutely suicidal, presenting to the adult emergency department with documented history of non-psychotic major depressive disorder.

Exclusion Criteria:

* Current psychotic or catatonic symptoms as determined by the hospital care team.
* Unable or unwilling to give consent for study participation (ability to provide consent will be established by treating physician)
* Lifetime DSM-V (medical history) diagnoses of schizophrenia, schizoaffective disorders, bipolar disorder, obsessive-compulsive disorder, and panic disorders.
* Meets current DSM-V substance use disorder of greater than mild severity (other than nicotine or marijuana)
* Significant pulmonary disease and/or requiring supplemental oxygen.
* Administration of other NMDA-receptor antagonist treatment (e.g., ketamine) within two weeks of entry into study.
* Contraindications for N2O (pneumothorax, bowel obstruction, middle ear occlusion, elevated intracranial pressure)
* Chronic cobalamin and/or folate deficiency treated with folic acid or vitamin B12.
* Women who are pregnant or breastfeeding
* Any other factor that in the investigators' judgment may affect patient safety or compliance.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-10-01 (Estimated); Primary Completion 2028-05-01 (Estimated); Study Completion 2028-10-01 (Estimated)

PRIMARY OUTCOMES:
Treatment Response Based on Changes in Computerized Adaptive Testing Scores | Up to 24-hours from baseline
  Monitor changes in Computerized Adaptive Testing Mental Health (CAT-MH) scores relating to suicide, depression, and anxiety; to determine whether a single 45-minute inhalation of nitrous oxide vs placebo reduces symptoms.
  The CAT-MH is a validated self-reporting electronic diagnostic that adaptively selects a small optimal set of items from a large bank of approximately 1,500 items, targeted to individuals current or historical level of severity and likelihood of 'suicide', 'depression', and 'anxiety'.
  Generated scores include severity and liklihood percentile:
  * suicide = (%) low, intermediate, high
  * depression = (%) normal, mild, moderate, severe
  * anxiety = (%) normal, mild, moderate, severe

SECONDARY OUTCOMES:
Treatment Compliance | Intervention completion, 45-minutes
  Evaluate compliance of an acutely suicidal population in an Emergency Department (ED) setting, to complete a single 45-minute inhalation of nitrous oxide vs placebo.
  Determined by 'ability', 'inability', or 'refusal' to complete the entire 45-minute inhalation session (nitrous oxide vs placebo).
Treatment Response Correlation to Lifetime Predictors Associated with Suicide | Up to 24-hours from baseline
  Evaluate if lifetime predictors (e.g., personal/family history of suicide attempts or suicide, history of alcohol dependence, and worst lifetime suicidal ideation) of eventual suicide correlate with the acute reduction in symptom severity following treatment.
  Lifetime predictors will be determined by medical and social history, and family history related to mental health.
  Symptom reduction is determined by changes in CAT-MH scores, over 24-hours from baseline.
  The CAT-MH is a validated self-reporting electronic diagnostic that adaptively selects a small optimal set of items from a large bank of approximately 1,500 items, targeted to individuals current or historical level of severity and likelihood of 'suicide', 'depression', and 'anxiety'.
  Generated scores include severity and liklihood percentile:
  * suicide = (%) low, intermediate, high
  * depression = (%) normal, mild, moderate, severe
  * anxiety = (%) normal, mild, moderate, severe
Rapid Treatment Response | At 30-minutes to 1-hour from intervention conclusion
  Evaluate any acute reduction in symptoms.
  Based on changes in CAT-MH scores (suicide, depression, anxiety) at 30-minutes to 1-hour following treatment. Study patients ability to complete self-administered CAT-MH following inhalation may impact time-point.
  The CAT-MH is a validated self-reporting electronic diagnostic that adaptively selects a small optimal set of items from a large bank of approximately 1,500 items, targeted to individuals current or historical level of severity and likelihood of 'suicide', 'depression', and 'anxiety'.
  Generated scores include severity and liklihood percentile:
  * suicide = (%) low, intermediate, high
  * depression = (%) normal, mild, moderate, severe
  * anxiety = (%) normal, mild, moderate, severe
Sustained Treatment Response | Up to 24-hours from intervention conclusion
  Evaluation of sustained response based on changes in CAT-MH scores at several time-points or until the patient is transferred or discharged from the ED.
  The CAT-MH is a validated self-reporting electronic diagnostic that adaptively selects a small optimal set of items from a large bank of approximately 1,500 items, targeted to individuals current or historical level of severity and likelihood of 'suicide', 'depression', and 'anxiety'.
  Generated scores include severity and liklihood percentile:
  * suicide = (%) low, intermediate, high
  * depression = (%) normal, mild, moderate, severe
  * anxiety = (%) normal, mild, moderate, severe

OTHER OUTCOMES:
Adverse Events | Through study completion, an average of 1-week
  Monitor adverse events and severity associated with study participation, including nausea and vomiting; or other symptoms determined 'probably', 'possibly', 'unrelated', or 'related' to the study intervention. This includes any unplanned escalation of care including pharmacological therapy for nausea, vomiting.
  Study patient safety is monitored by the investigators (MD) with experience in critical care anesthesia, as well as an experienced clinical research team responsible for data collection and reporting of events.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Nagele, MD, MSc, Principal Investigator — University of Chicago, Department of Anesthesia and Critical Care
Locations (1):
- University of Chicago Medicine, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No